CLINICAL TRIAL: NCT01165853
Title: Effects of Consuming Sugar-Sweetened Beverages With Meals for 10 Weeks on Hormones and Lipids
Brief Title: Effects of Consuming Sugar-Sweetened Beverages With Meals for 10 Weeks
Acronym: IPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 200412368; R01HL075675 (NIH)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Dyslipidemias | interventions — Glucose; Sugars; Fructose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucose (Other)
  Interventions: Other: Glucose
- Fructose (Other)
  Interventions: Other: Fructose

INTERVENTIONS:
Other: Glucose — 25% dose at 8-week intervention assigned to subjects.
  Other Names: sugar
  Arms: Glucose
Other: Fructose — 25% dose at 8-week intervention assigned to subjects.
  Other Names: sugar
  Arms: Fructose

SUMMARY:
The purpose of this study is compare the effects of consuming glucose- and fructose-sweetened beverages on appetite, body weight, body fat, and the amount of energy the body burns as well as effects on blood pressure, hormones, blood triglycerides and cholesterol, and the body's sensitivity to the insulin.

DETAILED DESCRIPTION:
The study is designed as a prospective, blinded diet intervention study during which the participants consume either fructose- or glucose-sweetened beverages (25% of energy) with meals. Experimental procedures, including 24-hour serial blood sampling, 26-h stable isotoped infusions, post-heparin blood collection, gluteal biopsies, metabolic rate monitoring, computed tomography scans of the abdomen, and Oral Glucose Tolerance and Disposal Tests, are performed during baseline and at the end of a 10-week intervention period at the UC Davis School of Medicine/Sacramento Veterans Affairs Medical Center Clinical Research Center (CCRC). During the 2-week inpatient baseline period, subjects are served energy balanced diets containing 15% of energy as protein, 30% as fat, and 55% as complex carbohydrate. Following the baseline period, the subjects reside at home for 8 weeks and consume their usual ad libitum diet along with 25% of energy requirements as fructose- or glucose-sweetened beverages. Subjects then return to the CCRC for the 2-week inpatient intervention period at the end of the study and are served energy-balanced diets containing 15% of energy as protein, 30% as fat, 30% as complex carbohydrate and 25% of energy as fructose- or glucose-sweetened beverage.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of stable body weight
* Women were post-menopausal based on a self-report of no menstruation for at least one year

Exclusion Criteria:

* evidence of diabetes
* renal or hepatic disease
* fasting serum TG concentrations >400 mg/dl
* hypertension (>140/90 mg Hg)
* surgery for weight loss
* individuals who smoked
* reported exercise of more than 3.5 hours/week at a level more vigorous than walking
* having used thyroid, lipid-lowering, glucose-lowering, anti-hypertensive, anti-depressant, or weight loss medications
* habitual ingestion of more than one sugar-sweetened beverage/day or more than two alcoholic beverages/day

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-07; Primary Completion 2007-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
24-hour triglyceride area under the curve | Baseline and 8-week intervention
  32 serial blood samples are collected over a 24 hour period.

SECONDARY OUTCOMES:
Insulin sensitivity index | Baseline and 8-week intervention
  Insulin sensitivity is assessed using the deuterated glucose disposal method.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Havel, D.V.M., Principal Investigator — University of California, Davis; Kimber L Stanhope, Ph.D, R.D., Study Director — University of California, Davis
Locations (1):
- Clinical Research Center, Sacramento, California, United States

REFERENCES:
- [Derived] Law HG, Stanhope KL, Zhang W, Myagmarsuren M, Jamshed ZM, Khan MA, Bang H, Havel PJ, Berglund L, Enkhmaa B. Lipoprotein(a) and diet: consuming sugar-sweetened beverages lowers lipoprotein(a) levels in obese and overweight adults. J Lipid Res. 2024 Aug;65(8):100588. doi: 10.1016/j.jlr.2024.100588. Epub 2024 Jul 4. PMID 38969065
- [Derived] Cox CL, Stanhope KL, Schwarz JM, Graham JL, Hatcher B, Griffen SC, Bremer AA, Berglund L, McGahan JP, Keim NL, Havel PJ. Circulating concentrations of monocyte chemoattractant protein-1, plasminogen activator inhibitor-1, and soluble leukocyte adhesion molecule-1 in overweight/obese men and women consuming fructose- or glucose-sweetened beverages for 10 weeks. J Clin Endocrinol Metab. 2011 Dec;96(12):E2034-8. doi: 10.1210/jc.2011-1050. Epub 2011 Sep 28. PMID 21956423
- [Derived] Stanhope KL, Griffen SC, Bremer AA, Vink RG, Schaefer EJ, Nakajima K, Schwarz JM, Beysen C, Berglund L, Keim NL, Havel PJ. Metabolic responses to prolonged consumption of glucose- and fructose-sweetened beverages are not associated with postprandial or 24-h glucose and insulin excursions. Am J Clin Nutr. 2011 Jul;94(1):112-9. doi: 10.3945/ajcn.110.002246. Epub 2011 May 25. PMID 21613559